CLINICAL TRIAL: NCT05673902
Title: An Open-Label Clinical Study of the Safety and Efficacy of RPH-104 in Preventing Recurrences in Patients With Idiopathic Recurrent Pericarditis
Brief Title: Study of the Safety and Efficacy of RPH-104 in Preventing Recurrences in Patients With Idiopathic Recurrent Pericarditis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: R-Pharm (Industry); Unimed Laboratories (Industry); Data Management 365 (Industry); Exacte Labs LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04018077
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Recurrent Pericarditis
Keywords: Pericarditis; Recurrent Pericarditis; RPH-104; subcutaneously
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RPH-104 80 mg (Experimental): RPH-104 80 mg SC once every 2 weeks for 24-60 weeks.
  (If the patient develops a pericarditis recurrence during the safety follow-up period, at the discretion of the investigator treatment with the study drug might be re-initiated according to the following regimen: a single dose of 160 mg SC (first injection) followed by a dose of 80 mg SC 7 days and 14 days after the first injection and at doses of 80 mg SC every two weeks thereafter.)
  Interventions: Biological: RPH-104

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Other Names: goflikicept; Arcerix

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of RPH-104 for long-term use in a population of patients with idiopathic recurrent pericarditis who completed the main study CL04018068.

The primary objective of the study is to evaluate the safety of RPH-104 80 mg once every 2 weeks in patients with idiopathic recurrent pericarditis who completed the main study.

DETAILED DESCRIPTION:
This long-term open-label study is an extension of the main double-blind, randomized, placebo-controlled study, CL04018068. This study will include the following periods:

* screening period - carried out on Day 0 (where Day 182, Week 26 from randomization in the main study CL04018068 will be considered as Day 0 of this study);
* re-screening period - up to 28 days (for patients who have completed the CL04018077 study);
* scheduled treatment period - 24-60 weeks (depends on the duration of treatment with RPH-104 during the main study CL04018068);
* safety follow-up period - 168 weeks. 60-week treatment re-initiation is possible in case of a disease recurrence reported during this period (with follow-up assessments 4 and 8 weeks after the last dosing of the investigational drug and telephone visits after 20, 32, 44, 56, 68, 80, 92 and 104 weeks after the administration of the final dose of the investigational drug, respectively).

It is planned that this study will include no more than 25 patients who completed the main study.

During the screening period, patients will be evaluated for eligibility for inclusion/non-inclusion in this study. Patients who do not meet these criteria will not receive treatment with the study drug.

Patients who meet the criteria for inclusion/non-inclusion in the study will enter the treatment period, where they will start open-label treatment with RPH-104 80 mg once every 2 weeks subcutaneously (SC).

The study drug to patients will be administered by qualified medical personnel every 2 weeks when the patient visits the study site, or at the patient's home by the patient him/herself. Safety and efficacy assessments are performed at Visit 1, Visit 2 (after 2 weeks) and then every 4 weeks according to the visits schedule.

After the patients receive the last dose of the study drug the treatment period will be considered completed and a 168 week period of safety follow-up will start. During this period, the patients will have to visit the study site after 4 weeks, then - after 8 weeks, and thereafter - every 12 weeks if in the Investigator's opinion it is considered safe and acceptable for a particular patient (it is possible to conduct the visits every 4 weeks until the completion of the study, if necessary in the Investigator's opinion and in agreement with Sponsor). There will also be eight telephone visits.

In case of a suspected recurrence of pericarditis, the patient will need to contact the study physician and come to the study site for an unscheduled visit. Recurrence of pericarditis is defined as the presence of at least two of the following symptoms in a patient:

* the chest pain intensity score according to the numeric rating scale (NRS) > 3 (in the absence of other possible reasons for the increase in the pain intensity);
* C-reactive protein (CRP) level > 5 mg/L (in the absence of other possible reasons for an increase in CRP levels);
* development of a new pericardial effusion or progression of the existing one in diastole according to echocardiography (EchoCG).

If recurrence of the disease is confirmed during the treatment period as well as if any of the above-described signs of relapse of pericarditis and its persistence (two consecutive visits) or a tendency to increase the values of the sign (estimated at two consecutive visits) are detected, therapy with the study drug could be canceled ahead of schedule or continued at a dose of 80 mg every 2 weeks with the addition of NSAIDs and / or colchicine at the discretion of the Investigator.

If the patient develops a pericarditis recurrence during the safety follow-up period, at the discretion of the investigator treatment with the study drug might be re-initiated in this patient for a duration of 60 weeks or therapy with alternative drugs of the researcher's choice might be prescribed (in this case, the patient will have to come to two follow-up visits - 4 and 8 weeks after the last dose of the study drug and perform eight telephone visits after 20, 32, 44, 56, 68, 80, 92 and 104 weeks after the administration of the last dose of the study drug. After that the patient will be considered to have completed the study). In case of study drug re-initiation, the drug will be administered according to the following regimen: a single dose of 160 mg (first injection) followed by a dose of 80 mg 7 days and 14 days after the first injection and at doses of 80 mg every two weeks thereafter (at the discretion of the investigator). At the discretion of the investigator, NSAIDs and/or colchicine might be used for the treatment of recurrences in these patients.

The assessment of the patient's condition will be carried out 3 days, 7 and 14 days, as well as 12 weeks after the continuation of the study therapy with the addition of NSAIDs and / or colchicine during the therapy period or after the study drug re-initiation during the safety monitoring period. The criterion for the resolution of the relapse is the presence of all the following signs simultaneously:

* the chest pain intensity score according to the numeric rating scale (NRS) ≤ 3 AND
* CRP level ≤ 5 mg/L AND
* absence or small (<10 mm) pericardial effusion or progression of the existing one in diastole according to echocardiography (EchoCG).

If the recurrence of the disease is resolved by the week 12, the patient will continue to use RPH-104 80 mg every 2 weeks and will conduct efficacy and safety assessments every 2 weeks for 12 weeks and thereafter every 4 weeks until the end of the scheduled treatment period or re-initiated therapy, depending on the period the study when the recurrence occurred. If glucocorticoid prescription is required by week 12 to resolve a recurrence, the investigated therapy will be canceled to the patient ahead of schedule.

If the patient develops a pericarditis recurrence after the study drug re-initiation (the patient already receives RPH-104 80 mg every 2 weeks during the safety monitoring period), as well as if any of the signs of a relapse of pericarditis and its persistence or a tendency to increase the values of the sign (as described above for the period of planned therapy), the use of RPH-104 might be canceled ahead of schedule or continued until the end of the period of re-initiated therapy at a dose of 80 mg every 2 weeks with the addition of NSAIDs and/or colchicine at the discretion of the investigator.

After the end of the re-initiated therapy, the patient will have to come to two follow-up visits - 4 or 8 weeks after the last dose of the study drug and perform eight telephone visits after 20, 32, 44, 56, 68, 80, 92 and 104 weeks after the administration of the last dose of the study drug.

No decrease or increase in the doses of the study drug (other than those described in this study) are envisaged in this study.

Patients who have discontinued the open-label therapy with the study drug early for any reason, should perform two safety follow-up visits at Week 4 and Week 8 after the last dose of the study drug and perform eight telephone visits after 20, 32, 44, 56, 68, 80, 92 and 104 weeks after the administration of the last dose of the study drug.

The duration of one patient participation in this open study is from 192 to 228 weeks, depends on the duration of the therapy period, which will be calculated for each patient, taking into account the duration of the RPH-104 use during the main study (CL04018068), as well as on the absence or presence of a pericarditis recurrence and the decision to resume the studied therapy in the safety follow-up period of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who fully completed per protocol a 24-week randomized withdrawal period (for the first 20 randomized patients), or the preparation therapy after the end of enrolment into the randomized withdrawal period in the main study CL04018068.

   OR Patient who fully completed per protocol the study CL04018077 (after repeated screening).
2. Voluntarily signed and dated Patient Informed Consent Form for participation in this study.
3. The patient's ability and willingness, according to the investigator, to follow the schedule of visits, the study procedures and follow the protocol requirements, including the following:

   * Come to the study site every 2 weeks for the study drug administration by qualified site staff; or
   * Learn how to perform subcutaneous injections and do it on their own at home as per protocol of this study.

Exclusion Criteria:

1. Unwillingness or inability of the patient to perform the study procedures in accordance with the Protocol.
2. Any medically important event that was reported in a patient during his/her participation in the main study CL04018068, and, in the opinion of the Investigator, is a reason for not including this patient in this open-label study.
3. Pregnant and lactating women or women planning pregnancy during the study or within 2 months after the last dose of the study drug.
4. Women of childbearing potential who do NOT agree to use highly effective contraception methods throughout the study, starting from the moment of signing the informed consent form and for at least 8 weeks after the last dose of the study drug.

   OR Men who are sexually active and do NOT agree to use highly effective contraception methods throughout the study, starting from the moment of signing the informed consent form and for at least 8 weeks after the last dose of the study drug.

   Highly effective contraception methods include:
   * sterilization in women: surgical bilateral removal of the ovaries (with or without removal of the uterus) or ligation of the fallopian tubes at least 6 weeks before the start of the study therapy. In the case of removal of only the ovaries, the reproductive status of a woman should be confirmed by a subsequent assessment of hormone level;
   * sterilization in men, at least 6 months before the start of the study therapy with proper documentation of the absence of sperm in the ejaculate after vasectomy. For women participating in the study, a sexual partner after a vasectomy should be the only partner;
   * using a combination of any two of the following methods (a+b or a+c or b+c):

     1. oral, injectable or implanted hormonal contraceptives; in the case of the use of oral contraceptives, women should continuously use the same drug for at least 3 months before the start of the study therapy;
     2. an intrauterine device or contraceptive system;
     3. barrier methods of contraception: condom or occlusive cap (diaphragm or cervical cap/contraceptive vaginal ring) with spermicidal foam/gel/film/cream/vaginal suppository.
5. The need to use a live (attenuated) vaccine during the study or within 3 months after the last dose of the study drug. Live attenuated vaccines include vaccines against the following viruses: measles, rubella, mumps, chickenpox, rotavirus, flu (as a nasal spray), yellow fever, polio (oral polio vaccine); vaccines against tuberculosis (BCG), typhoid fever (oral typhoid vaccine) and typhus (typhus vaccine). Immunocompetent family members of the patient should not be vaccinated with the oral polio vaccine during the patient's participation in the study.
6. Other medical conditions or laboratory abnormalities, which may increase the potential risk associated with participation in the study and treatment with the study drug, or may affect the interpretation of the results of the study, and which, in the opinion of the Investigator lead to patient ineligibility for this study.
7. Parallel participation in other clinical trials (except for the main study CL04018068) at the time of screening or the use of any unapproved (investigational) drugs (except for RPH-104) less than 4 weeks or 5 half-lives (whichever is greater) before screening.

   For patients undergoing repeated screening, the following criteria are additionally applicable:
8. Hypersensitivity to the test drug (RPH-104), and/or its components /excipients and/or drugs of the same chemical class.
9. Previous use of drugs:

   * rilonacept - less than 6 weeks before the initial assessment (the day of the re-screening visit),
   * kanakinumab - less than 12 weeks before the initial assessment (the day of the re-screening visit),
   * anakinra - less than 5 days before the initial assessment (the day of the re-screening visit),
   * drugs of the TNF inhibitor class, IL-6 inhibitors, janus kinase inhibitors - less than 12 weeks before the initial assessment (the day of the re-screening visit),- - immunosuppressants (azathioprine, cyclosoprine, mycophenolate, mofetil, tacrolimus, sirolimus, mercaptopurine) - less than 24 weeks before the initial assessment (the day of the re-screening visit),
   * methotrexate - less than 2 weeks before the initial assessment (the day of the re-screening visit),
   * any other biological drugs in less than 5 periods half-life before the start of therapy.
10. Any conditions or signs in the patient that, according to the investigator's judgement, indicate a disorder (suppression) of the patient's immune response and/or significantly increase the risk of immunomodulatory therapy, including, but not limited to, the following:

    * active bacterial, fungal, viral or protozoal infection revealed at the beginning of the screening period;
    * opportunistic infections and/or Kaposi's sarcoma at the beginning of the screening period;
    * chronic bacterial, fungal or viral infection requiring systemic therapy at the beginning of the screening period;
    * HIV-infection, hepatitis B or C (patients with treated hepatitis C and negative polymerase chain reaction (PCR) tests after 3 and 6 months are regarded as cured from hepatitis C and can be included in this study);
11. A history of active tuberculosis or the presence of risk factors or signs indicating the presence of active or latent infection caused by M. Tuberculosis, including but not limited to the following:

    * living in specific conditions that increase the risk of contacts with tuberculosis-infected patients, such as prisons, gathering of homeless people etc. over the past year until the beginning of the main treatment period;
    * occupational exposure at a medical institution in the settings of unprotected contact with patients with a high risk of tuberculosis or patients with tuberculosis during the last year before the start of the screening period;
    * close contact, i.e. being in the same room (at home or in another confined environment) for an extended period of time (days or weeks rather than minutes or hours) with a person with active pulmonary tuberculosis within the past year prior to the beginning of the treatment period;
    * test results indicating active tuberculosis or latent infection caused by M. Tuberculosis: positive result of QuantiFERON-TB/T-SPOT test.TB during the screening period; findings of chest X-ray exam in two views confirming pulmonary tuberculosis during the screening period.
12. History of alcohol abuse or psychoactive substances abuse as assessed by the Investigator.
13. Severe renal impairment: creatinine clearance by Cockcroft-Gault formula <30 mL/min at the screening.
14. Presence of any of the following at the screening:

    * absolute neutrophil count <1.5 х 10^9/L,
    * white blood cells (WBC) count <3.5 х 10^9/L,
    * platelet count <100 х 10^9/L,
    * hemoglobin ≤ 80 g/L,
    * glycated hemoglobin (HbA1c) ≥ 8% (to be evaluated only in patients with diabetes mellitus),
    * alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 3.0 х upper limit of normal (ULN),
    * total bilirubin >1.5 х ULN (except for cases of documented Gilbert's syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs), by System Organ Class and Preferred Term | Up to week 228
Incidence of Treatment-Emergent Serious Adverse Events (SAEs), by System Organ Class and Preferred Term | Up to week 228
Incidence of Treatment-Emergent Adverse Events of Special Interest (AESI), by System Organ Class and Preferred Term | Up to week 228
Incidence rate for serious adverse events (SAEs) | Up to week 228
  Incidence rate, expressed as the number of events per 100 patient-years of follow-up, for SAEs
Incidence rate for adverse events of special Interest (AESI) | Up to week 228
  Incidence rate, expressed as the number of events per 100 patient-years of follow-up, for AESI

SECONDARY OUTCOMES:
Proportion of patients with pericarditis recurrence during 24 weeks of therapy in the study and during the entire period of the study treatment | weeks 24, 60
  The criterion for the development of disease recurrence is the appearance of at least two of the following signs:
  * the chest pain intensity scores according to the numeric rating scale (NRS) > 3 (in the absence of other possible reasons for the increase in the pain intensity);
  * CRP level > 5 mg/L (in the absence of other possible reasons for an increase in CRP levels);
  * development of a new pericardial effusion or progression of the existing one in diastole according to EchoCG.
  NRS contains 11 values from 0 to 10 points, where 0 is no pain, 10 is unbearable pain.
Proportion of patients with pericarditis recurrence during 24 weeks of the follow-up period and during the entire follow-up period of the study | weeks 24, 228
  The criterion for the development of disease recurrence is the appearance of at least two of the following signs:
  * the chest pain intensity scores according to the NRS> 3 (in the absence of other possible reasons for the increase in the pain intensity);
  * CRP level > 5 mg/L (in the absence of other possible reasons for an increase in CRP levels);
  * development of a new pericardial effusion or progression of the existing one in diastole according to EchoCG.
  NRS contains 11 values from 0 to 10 points, where 0 is no pain, 10 is unbearable pain.
Change from the baseline in the chest pain intensity as assessed by patients on the numeric rating scale during a 24-week treatment period and the entire study treatment period | baseline, weeks 24, 60
  Change from the baseline (i.e. the last available measurement before the first dose of the study drug in the main study CL04018068) in the chest pain intensity as assessed by patients on the numeric rating scale (NRS) during a 24-week treatment period and the entire study treatment period.
  NRS contains 11 values from 0 to 10 points, where 0 is no pain, 10 is unbearable pain.
Change from the baseline in patients' overall health scores on the numeric rating scale period during a 24-week treatment period and the entire study treatment period. | baseline, weeks 24, 60
  The patient's overall health will be assessed using a NRS containing 11 values from 0 to 10 points, where 0 is very good, 10 is very poor.
Change from the baseline in the physician's overall disease score on the numeric rating scale period during a 24-week treatment period and the entire study treatment period | baseline, weeks 24, 60
  Global disease activity is assessed by the physician using a NRS containing 11 values from 0 to 10 points, where 0 is the absence of active disease, 10 is the maximum activity of the disease.
Change from the baseline in C-reactive protein (CRP) levels during 24 weeks of therapy in the study and during the entire period of the study treatment | baseline, weeks 24, 60
Change from the baseline in the size of pericardial effusion according to Echo-CG during 24 weeks of therapy in the study and during the entire period of the study treatment | baseline, weeks 24, 60
Change from the baseline in the patient quality of life as assessed using the SF-36 questionnaire period during a 24-week treatment period and the entire study treatment period | baseline, weeks 24, 60
  Change from the baseline in the patient quality of life as assessed using the SF-36 questionnaire during the study treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (1):
- National medical research center named after V. A. Almazov, Saint Petersburg, Russia